CLINICAL TRIAL: NCT05836883
Title: A Phase IB/IIA Study of ExoFlo, an Ex Vivo Culture-expanded Adult Allogeneic Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicle Isolate Product, for the Treatment of Perianal Fistulizing Crohn's Disease
Brief Title: Study of ExoFlo for the Treatment of Perianal Fistulas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges.
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DB-EF-PFCD-1a
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Perianal Fistula; Crohn's Disease
Keywords: Perianal Fistula; Perianal Fistulizing Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Multicenter, Placebo-controlled, Dose-escalation Design, Randomized Controlled Trial.
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1: Placebo (Placebo Comparator): Local injection 15 mL of normal saline on Day 0
  Interventions: Other: Local injection of normal saline
- Cohort 2: Placebo (Placebo Comparator): Local injection 30 mL of normal saline on Day 0
  Interventions: Other: Local injection of normal saline
- Cohort 3: Placebo (Placebo Comparator): Local injection 30 mL of normal saline on Day 0 and Month 3
  Interventions: Other: Local injection of normal saline
- Cohort 1: Treatment (Experimental): Local injection of 15 mL of ExoFlo on Day 0
  Interventions: Biological: ExoFlo
- Cohort 2: Treatment (Experimental): Local injection of 30 mL of ExoFlo on Day 0
  Interventions: Biological: ExoFlo
- Cohort 3: Treatment (Experimental): Local injection of 30 mL of ExoFlo on Day 0 and Month 3
  Interventions: Biological: ExoFlo

INTERVENTIONS:
Biological: ExoFlo — Local injection of bone marrow mesenchymal stem cell derived extracellular vesicles
  Arms: Cohort 1: Treatment; Cohort 2: Treatment; Cohort 3: Treatment
Other: Local injection of normal saline — Placebo
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo

SUMMARY:
To evaluate the safety and feasibility of ExoFlo as a treatment for Perianal Fistulizing Crohn's Disease.

DETAILED DESCRIPTION:
This is a phase IB/IIA, multicenter, single-blind, placebo-controlled, dose-escalation design, randomized controlled trial for the treatment of Perianal Fistulizing Crohn's Disease.

Subjects will be randomized 2:1 Investigational Medicinal Product (IMP) to normal saline (NS) in 3 cohorts of 12 subjects as follows:

Cohort 1: Local injection of 15 mL of IMP or NS on Day 0 (8 IMP, 4 NS) Cohort 2: Local injection of 30 mL of IMP or NS on Day 0 (8 IMP, 4 NS) Cohort 3: Local injection of 30 mL of IMP or NS on Day 0 and Month 3 (8 IMP, 4 NS)

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women 18-75 years of age with a diagnosis of Crohn's Disease (CD) for at least six months duration.
2. Single and/or Multi-tract Perianal fistula(s).
3. Failed at least one medical therapy within the last year including, but not limited to, antibiotics, immunomodulators (6-MP, methotrexate, azathioprine), monoclonal antibodies (infliximab, adalimumab, certolizumab, ustekinumab, golimumab, vedolizumab), or small molecule inhibitors.
4. Previous failed surgical intervention, including seton placement at least two weeks prior, or are not candidates for surgical intervention or are not willing to undergo surgical intervention for the management of their fistula.
5. Medical therapy for CD stable for at least 2 months prior to administration of IMP. Changes in dosing or dosing intervals related to serum drug levels are permitted.
6. Ability to comply with protocol.
7. Competent and able to provide written informed consent.

Exclusion Criteria:

1. Active perianal abscess or infection at the time of screening, enrollment, or at the time of investigational product administration
2. Clinically significant medical conditions within the six months before administration of IMP that would, in the opinion of the investigators, compromise the safety of the subject.
3. History of cancer including melanoma (with the exception of localized skin cancers) within one year of screening.
4. History of colorectal cancer within 2 years
5. Subjects who have a diagnosis of coagulation disorders and/or are currently on anti-coagulant therapy
6. Investigational drug within one month of treatment
7. Pregnant or breast feeding or trying to become pregnant.
8. Presence of a rectovaginal fistula
9. Presence of an ileal anal pouch and/or history of proctectomy
10. The presence of severe proctitis
11. Any condition which, in the opinion of the investigator, would make it unsafe or unsuitable for patients to undergo Magnetic Resonance (MR) evaluations (i.e., presence of implantable or external MR unsafe device that cannot be removed, body weight exceeding limitations, claustrophobia etc.).
12. A participant who is unwilling to use medically acceptable contraception methods during participation in study
13. The following out of range laboratory results at screening (result may be repeated)

    * WBC >11 x 109 /L
    * Hemoglobin < 8 g/dl
    * Platelet count <100,000/mL
    * AST/ALT >2 times the upper limit of normal
    * Creatinine >2 umol/L
    * PT/INR: outside normal limits
    * Hemoglobin A1c>6.5 mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility | 12 Months
  Safety will be defined as the rate of Adverse Events (AEs) or Severe Adverse Events (SAEs) related to IMP and administration of IMP in this patient population. Safety and feasibility will be evaluated for one dose of 15 mL or 30 mL ExoFlo or two doses of 30 mL ExoFlo in subjects with perianal fistula(s) in the setting of Crohn's Disease.

SECONDARY OUTCOMES:
Healing | 12 Months
  To evaluate the efficacy for one dose of 15 mL or 30 mL ExoFlo or two doses of 30 mL ExoFlo in subjects with perianal fistula(s) in the setting of Crohn's Disease. Subjects will be evaluated for healing progress: complete healing, partial healing, lack of response, or treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC
Locations (1):
- Direct Biologics Investigational Site, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Direct Biologics, LLC — https://directbiologics.com/